CLINICAL TRIAL: NCT01076101
Title: Mapping Autoimmune Phenotypes in Multiplex Families (MADGC 2)
Brief Title: Autoimmunity in Sisters of Lupus Patients
Acronym: SisSLE
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter Gregersen, Principal Investigator, Northwell Health
Other Study IDs: 09-263; R01AI068759 (NIH)
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; sister; autoimmune disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — We will use your DNA blood sample to study the function of genes and biomarkers and gain understanding of their role in protection against disease or the role they play in increasing the risk factors of developing lupus. No, you will not get test results since the information we gather is only useful for research and is not diagnostic. Participation in this study is not a substitute for regular medical care.
  The information and blood sample that is collected for research will be analyzed for many years and it is not possible to know how long this analysis and follow-up will take. Therefore, participation allows the information and banking of your blood sample to be indefinite.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sisters who have a diagnosis of SLE: Sisters who have a diagnosis of SLE
- Unaffected Sisters: Sisters of SLE patients who do not have a diagnosis of SLE

SUMMARY:
This study enrolled over 400 unaffected sisters of young women diagnosed with SLE. These unaffected sisters are being followed with an annual health questionnaire (CSQ) and blood sample.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease that causes inflammation and is accompanied by the development of autoantibodies. The inflammation caused by SLE may affect the skin, joints, lungs, blood, kidneys and nervous system. The cause of SLE is unknown, but research has indicated that it is caused by a combination of genetic and environmental factors.

Autoimmune diseases often run in families. Close relatives of people with these diseases are at greater risk of developing the same or another autoimmune disease. The study is designed to determine several things: If sisters of people with SLE make the same antibodies that are present in people with SLE, whether or not environmental factors affect the chances of developing these antibodies and if so what these environmental factors may be, if the presence of these antibodies in healthy people leads to increased risk for the development of SLE.

This study enrolled over 400 unaffected sisters of young women diagnosed with SLE. These unaffected sisters are being followed with an annual health questionnaire (CSQ) and blood sample.

Participation is voluntary and participants can stop participating at any time.

ELIGIBILITY:
Sister Diagnosed with SLE:

Inclusion Criteria:

1. Proband must be a female and have documented SLE that meets ACR criteria. SLE must be diagnosed by and including age 40.
2. Proband must have at least one biological sister ≥ 10 years of age and ≤ 45 who is available and willing to donate a blood sample and enroll in a longitudinal study. Both full and half siblings qualify.

Exclusion Criteria:

If inclusion criteria above are met for the proband, there are no exclusions.

Sister who does not have SLE:

Inclusion Criteria:

1. Female with a full or half sister who has been documented SLE that meets ACR criteria.
2. Sister must be currently between ages ≥ 10 and ≤ 45 at the time of enrollment and not have a diagnosis of SLE.
3. Sister must be able to complete questionnaires and should be willing to donate a blood sample at baseline and follow-up.
4. Sister should communicate to the recruiter that she is willing to be followed for a period of at least two years by phone and/or internet.

Exclusion Criteria:

If Sister meets inclusion criteria, there will be no exclusions.

Ages: 10 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sisters: One sister must be diagnosed with Systemic Lupus Erythematous ( SLE ) by and including age 40 who has a sister(s) or half sister(s) not affected with SLE currently between the ages of 10 and 45 are being recruited nation wide through community and physician referrals.
Sampling Method: Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2009-02; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
To identify biomarkers that can predict the future development of clinical disease in subjects at risk, or alternatively, indicate that progression to overt clinical disease is unlikely | 5 years

SECONDARY OUTCOMES:
To understand the preclinical biological and immunological events that precede the development of systemic lupus | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter K Gregersen, MD, Principal Investigator — NorthShore -LIJ The Feinstein Institute for Medical Research
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No